CLINICAL TRIAL: NCT03420053
Title: Clinical Trial to Evaluate the Safety, Immunogenicity and Efficacy of Direct Venous Inoculation of Plasmodium Falciparum Sporozoite Vaccine (PfSPZ Vaccine) in HIV Negative and HIV Positive Tanzanian Adults
Brief Title: Study to Evaluate Safety, Immunogenicity and Efficacy of PfSPZ Vaccine in HIV Negative and HIV Positive Tanzanian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Medical Care Development, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BSPZV3a
Record Dates: First submitted 2017-12-13; First posted 2018-02-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Malaria; Malaria,Falciparum
Keywords: PfSPZ Vaccine; HIV+; Plasmodium falciparum; Sporozoites
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 HIV- vaccine recipients (Experimental): Group 1: n=6, HIV negative vaccine recipients will receive 9.0x10^5 PfSPZ Vaccine at 0, +2, +4, +6 and +28 days. Total no. of volunteers in Group 1, n=9, where volunteers will be randomized in a 1:2 ratio to receive either normal saline placebo (NS) or PfSPZ Vaccine.
  Efficacy will be assessed by controlled human malaria infection (CHMI) at +3 weeks (+2 to +10 weeks) after the last dose of PfSPZ Vaccine. CHMI will be by DVI of 3,200 PfSPZ Challenge.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge
- Group 1 HIV- NS controls (Placebo Comparator): Group 1: n=3, HIV negative NS placebo recipients will receive NS at 0, +2, +4, +6 and +28 days. Total no. of volunteers in Group 1, n=9, where volunteers will be randomized in a 1:2 ratio to receive either NS placebo or PfSPZ Vaccine.
  Efficacy will be assessed by CHMI at +3 weeks (+2 to +10 weeks) after the last dose of NS. CHMI will be by DVI of 3,200 PfSPZ Challenge.
  Interventions: Other: Normal Saline Placebo; Biological: PfSPZ Challenge
- Group 2a HIV+ vaccine sentinels (Experimental): Group 2a: n=3, HIV positive vaccine recipients will receive 4.5x10^5 PfSPZ Vaccine at 0, +2, +4, +6 and +28 days.
  Interventions: Biological: PfSPZ Vaccine
- Group 2b HIV+ vaccine recipients (Experimental): Group 2b: n=6, HIV positive vaccine recipients will receive 9.0x10^5 PfSPZ Vaccine at 0, +2, +4, +6 and +28 days. Total no. of volunteers in Group 2b, n=9, where volunteers will be randomized in a 1:2 ratio to receive either NS placebo or PfSPZ Vaccine.
  Efficacy will be assessed by CHMI at +3 weeks (+2 to +10 weeks) after the last dose of PfSPZ Vaccine. CHMI will be by DVI of 3,200 PfSPZ Challenge.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge
- Group 2b HIV+ placebo controls (Placebo Comparator): Group 2b: n=3, HIV positive NS placebo recipients will receive NS at 0, +2, +4, +6 and +28 days. Total no. of volunteers in Group 2b, n=9, where volunteers will be randomized in a 1:2 ratio to receive either NS placebo or PfSPZ Vaccine.
  Efficacy will be assessed by CHMI at +3 weeks (+2 to +10 weeks) after the last dose of NS. CHMI will be by DVI of 3,200 PfSPZ Challenge.
  Interventions: Other: Normal Saline Placebo; Biological: PfSPZ Challenge

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, metabolically active, non-replicating, radiation-attenuated, cryopreserved Pf sporozoites.
  Arms: Group 1 HIV- vaccine recipients; Group 2a HIV+ vaccine sentinels; Group 2b HIV+ vaccine recipients
Other: Normal Saline Placebo — 0.9% sodium chloride solution
  Arms: Group 1 HIV- NS controls; Group 2b HIV+ placebo controls
Biological: PfSPZ Challenge — Aseptic, purified, live, infectious, cryopreserved Pf sporozoites.
  Arms: Group 1 HIV- NS controls; Group 1 HIV- vaccine recipients; Group 2b HIV+ placebo controls; Group 2b HIV+ vaccine recipients

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to evaluate safety and tolerability of PfSPZ Vaccine administered as five doses of 9.0x10^5 PfSPZ or normal saline at 0, +2, +4, +6 and +28 days to healthy HIV negative adult volunteers and healthy HIV positive volunteers in Tanzania.

DETAILED DESCRIPTION:
This trial is a single center trial designed to assess the safety, tolerability, immunogenicity and efficacy of PfSPZ Vaccine (9.0x10^5 PfSPZ given at 0, +2, +4, +6 and +28 days (Group 1, HIV negative, and Group 2, HIV positive)). Controls will receive parallel injections with normal saline (NS). All administrations of PfSPZ or NS will be by direct venous inoculation (DVI).

Twenty-one male and female adult volunteers, aged from 18 to 45 years, who live in and around the Bagamoyo township, will be enrolled based on pre-defined inclusion and exclusion criteria. 12/21 subjects will be HIV positive volunteers (who clinical stage 1) on stable anti-retroviral therapy (ART) for at least 3 months with a CD4+ cell count above 500 cells/μL at screening. The rest (9/21) will be healthy HIV negative adults.

Treatment allocation will be double-blind within Group 1 and 2b but not between the groups or subgroups. Immunizations will begin with healthy HIV negative volunteers first (Group 1), before inoculation of HIV positive volunteers (Groups 2a and 2b). Transitioning from immunization of HIV negative to immunization of HIV positive will begin by immunizing a sentinel group of 3 HIV positive individuals with a reduced vaccine dose of 4.5x10^5 PfSPZ (Group 2a). This transition will be staggered by at least two (2) weeks, to allow for a safety data review. If the safety data do not meet pause criteria, this will signal a "go" for transitioning to immunizations of sentinel group of three (3) HIV positive volunteers. If pause criteria are met, there will be no immediate transition, and instead an ad-hoc meeting of the Safety Monitoring Committee (SMC) will be called for an independent review and recommendation. Transition from the unblinded HIV positive sentinel Group 2a to the full study cohort of double blinded placebo controlled HIV positive volunteers (Group 2b), will also be staggered for at least two (2) weeks. There will be a scheduled review by the SMC of safety data collected from the sentinel HIV positive group for up to 7 days after the fourth immunization. After the safety review, transition to the main HIV positive group (Group 2b) will take into account the SMC recommendation(s).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, from 18 to 45 years of age
* Long term (at least two years) or permanent residence in the Bagamoyo district or nearby districts in Coastal and Dar-es-Salaam regions
* Availability through mobile phone 24 hours a day during the whole study period
* Ability and willingness to complete the study visit schedule for safety follow-up and protocol compliance
* Agreement to provide personal contact information and contact information of a third party household member or close friend to study team
* Agreement not to participate in any other clinical study involving investigational medicinal products during the study period, except enrollment in observational studies (such a co-enrollment must be approved by the PI)
* Agreement to release medical and other information concerning contra-indications for participation in the study, and to be attended by a study clinician for physical examination and clinical investigations including electrocardiogram (ECG)
* Willingness to undergo all blood, urine and stool tests (as specified in the protocol) and additional tests that may be ordered by the study clinician to rule-out significant abnormality(ies)
* Female volunteers must be willing to take measures not to become pregnant if selected for participation in the trial and to undergo serum pregnancy test at screening and at defined time-points during the trial
* Volunteers for enrollment into HIV positive sub-groups must have:

  1. Documented HIV infection, be in general good health and on stable ART use for at least three (3) months, preferably six (6), prior to screening
  2. WHO clinical stage 1 of HIV disease
  3. CD4+ T-cell count >500 cells/μL at screening
  4. Attending a care and treatment centre (CTC) within the study area for medical management of HIV infection, and agreeing to maintain regular attendance to such care and treatment centre while participating in the study
  5. Agreement to allow the clinical team to contact and coordinate care with the volunteer's HIV CTC.
* Correctly answering 10 out of 10 questions during informed consent process to demonstrate the understanding of study design, study procedures, risks and benefits
* Signing and dating written informed consent, in accordance with local practice.

Exclusion Criteria:

* Previous receipt of an investigational malaria vaccine or drug in the last 5 years
* Receipt of standard vaccinations within 4 weeks prior to the first immunization with a PfSPZ product or are planning to take standard vaccinations during the trial through 4 weeks following the last injection with a PfSPZ product
* Participation in any other clinical trial involving investigational medicinal products within 30 days prior to the onset of the study
* Clinically significant cardiac abnormalities as indicated by history, physical examination or clinically significant abnormalities in electrocardiogram (ECG)
* Positive family history in a 1st or 2nd degree relative for cardiac disease at age< 50 years old
* A history of psychiatric disease
* History of afebrile seizures, atypical febrile seizures or epilepsy
* History of drug or alcohol abuse interfering with normal social function
* History of chronic immunodeficiency condition (other than HIV) or autoimmune disease
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months prior to study onset (ART and inhaled and topical corticosteroids are allowed)
* Meeting exclusion criteria based on the protocol algorithm for assessment of TB disease risk
* Currently on Co-Trimoxazole (trimethoprim/sulfamethoxazole) prophylactic treatment (CPT)
* Currently taking rifampin (isoniazid is not an exclusion criterion)
* Body mass index (BMI) of <18 or >30 Kg/m2
* Females who are pregnant (as indicated by positive serum pregnancy test), nursing, or plan on becoming pregnant or nurse within the duration of trial
* Newly diagnosed with positive HIV infection at screening
* Positive hepatitis (B or C virus) tests
* Symptoms, physical signs and laboratory values suggestive of clinically significant systemic disorders or any other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Medical, social condition or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation, may impair the volunteer's ability to give informed consent or effectively participate in the study, may significantly increase the risk to the volunteer because of participation in the study or may impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Safety of PfSPZ Vaccine - solicited symptoms | From day of vaccination to 7-days post vaccination.
  Occurrence of solicited symptoms during a 7-day surveillance period after vaccination (day of vaccination (Vx) and +7 days post vaccination).
Safety of PfSPZ Vaccine - unsolicited symptoms | From day of vaccination to 28-days post vaccination.
  Occurrence of unsolicited symptoms during a 28-day surveillance period after each vaccination.
Safety of PfSPZ Vaccine - laboratory abnormalities | Day of immunization to approximately 11 weeks after the last vaccination (approximately 36 weeks).
  Occurrence of laboratory abnormalities including significant drops in CD4 T cell counts or increases in viral load.
Safety of PfSPZ Vaccine - serious adverse events | Day of immunization to approximately 11 weeks after the last vaccination (approximately 36 weeks).
  Occurrence of serious adverse events during the study period.
Safety of PfSPZ Vaccine - breakthrough infection | Day of immunization to approximately 11 weeks after the last vaccination (approximately 36 weeks).
  - Occurrence of Pf infection of vaccine type detected at any point after the first vaccination (retrospectively determined).

CONTACTS AND LOCATIONS:
Overall Officials: Said Jongo, MD, MMED, Principal Investigator — Ifakara Health Institute
Locations (1):
- Bagamoyo Research and Training Center of the Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Jongo S, Church LWP, Milando F, Qassim M, Schindler T, Rashid M, Tumbo A, Nyaulingo G, Bakari BM, Athuman Mbaga T, Mohamed L, Kassimu K, Simon BS, Mpina M, Zaidi I, Duffy PE, Swanson PA 2nd, Seder R, Herman JD, Mendu M, Zur Y, Alter G, Kc N, Riyahi P, Abebe Y, Murshedkar T, James ER, Billingsley PF, Sim BKL, Richie TL, Daubenberger C, Abdulla S, Hoffman SL. Safety and protective efficacy of PfSPZ Vaccine administered to HIV-negative and -positive Tanzanian adults. J Clin Invest. 2024 Jan 9;134(6):e169060. doi: 10.1172/JCI169060. PMID 38194272